CLINICAL TRIAL: NCT01033045
Title: Epidemiological Study to Evaluate the Management of Patients With Chronic Hepatitis C and Previous Treatment Failure
Status: Completed | Type: Observational
Sponsor: Fundacion IMIM (Other)
Responsible Party: Principal Investigator, Ricard Sola, MD, Fundacion IMIM
Other Study IDs: AGORA
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Viral; Non-A; Non-B; Parenterally-Transmitted
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe the management of patients with chronic hepatitis C and previous treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 18 years old.
* Patients with hepatitis C who had previously failed to the standard therapy.
* Patients who have given written informed consent to participate in the study.

Exclusion Criteria:

* Patients with clinical and/or social conditions that might interfere with the development of the study (terminal diseases, cognitive detriment, severe psychiatric disease which prevent from obtaining the information required, prolonged absences during the study).
* Patients who are participating in other research trials or under treatment with any agent contraindicated according to the summary of product characteristics or other circumstance which requires a patient management different from the investigator's regular clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes older than 18 years old with hepatitis C who had previously failed to the standard therapy.
Sampling Method: Probability Sample
Enrollment: 2178 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Describe the management of patients with chronic hepatitis C and previous treatment failure | 6 years

SECONDARY OUTCOMES:
To know the frequency of the causes for not responding to the previous treatment: lack of adherence to treatment, incomplete dose of antiviral treatment, insufficient treatment duration or treatment resistance. | 6 years
To assess the percentage of patients with previous treatment failure who are not candidates for re-treatment and its causes. | 6 years
To evaluate the implementation of current recommendations based on the cause of the previous therapeutic failure, in patients with chronic hepatitis C in whom a new course of the antiviral treatment is decided to be administered. | 6 years
To know the causes of the dose modifications and withdrawal of treatment during the follow-up period in patients who start re-treatment. | 6 years
To know the percentage of patients that achieve sustained viral response when implementing the recommendations based on the cause of the previous therapeutic failure. | 6 years
To determine the presence of the polymorphism rs12979860 in the gene IL 28B located on chromosome 19. | 6
  The rs12979860 polymorphism in the gene IL 28B that is located on chromosome 19 showed to be strongly associated with the development of sustained viral response (SVR) in patients with chronic hepatitis C treated with PEG-IFN-α/RBV. Patients with this polymorphism clear the virus more easily.
Compare the management of patients with chronic hepatitis C prior treatment failure before and after the appearance of new treatments. | 3

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Solà Lamoglia, Dr., Principal Investigator — Hospital del Mar; Ramón Planas Vila, Dr., Principal Investigator — Hospital Germans Tries i Pujol, Barcelona; Javier García-Samaniego, Dr., Principal Investigator — Hospital Carlos III, Madrid; Moisés Diago, Dr., Principal Investigator — Hospital General Universitario de Valencia; Manuel Romero, Dr., Principal Investigator — Hospital de Valme, Sevilla; José Luís Calleja, Dr, Principal Investigator — Hospital Puerta del Hierro, Madrid
Locations (104):
- Spain (104):
  - H. de Antequera, Antequera, Andalusia
  - H. Puerta de Mar, Cadiz, Andalusia
  - H. Puerto Real, Cadiz, Andalusia
  - H. Vírgen de las Nieves, Granada, Andalusia
  - H. Infanta Elena, Huelva, Andalusia
  - H. de Jaen, Jaén, Andalusia
  - H. de Jerez, Jerez de la Frontera, Andalusia
  - H. Carlos Haya, Málaga, Andalusia
  - H. Vírgen de la Victoria, Málaga, Andalusia
  - H. de Valme, Seville, Andalusia
  - H. San Jorge, Huesca, Aragon
  - H. Clínico de Zaragoza, Zaragoza, Aragon
  - H. Miquel Servet, Zaragoza, Aragon
  - H. Son Dureta, Mallorca, Balearic Islands
  - H. Son Llàtzer, Mallorca, Balearic Islands
  - H. Manacor, Manacor, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - H. Basurto, Bilbao, Basque Country
  - H. de Galdakano, Bilbao, Basque Country
  - H. las Cruces, Bilbao, Basque Country
  - H. de Donosti, Donostia / San Sebastian, Basque Country
  - H. Carlos III, Madrid, C de Madrid
  - H. de Henares, Alcalá de Henares, C. de Madrid
  - Fundación de Alcorcón, Alcorcón, C. de Madrid
  - H. de Getafe, Getafe, C. de Madrid
  - H. 12 de Octubre, Madrid, C. de Madrid
  - H. Fundación Jiménez Díaz, Madrid, C. de Madrid
  - H. la Paz, Madrid, C. de Madrid
  - H. la Princesa, Madrid, C. de Madrid
  - H. Príncipe de Astúrias, Madrid, C. de Madrid
  - H. Severo Ochoa, Madrid, C. de Madrid
  - H. de Móstoles, Móstoles, C. de Madrid
  - H. Infanta Cristina, Parla, C. de Madrid
  - H. Infanta Sofía, San Sebastián de los Reyes, C. de Madrid
  - H. de Alcoy, Alcoy, C. Valenciana
  - H. General de Alicante, Alicante, C. Valenciana
  - H. Marina Baixa, Alicante, C. Valenciana
  - H. de Castellón, Castellon, C. Valenciana
  - H. de Elche, Elche, C. Valenciana
  - H. Vega Baja, Orihuela, C. Valenciana
  - H. Clínico de Valencia, Valencia, C. Valenciana
  - H. General de Valencia, Valencia, C. Valenciana
  - H. de Xàtiva, Xàtiva, C. Valenciana
  - H. Insular, Gran Canaria, Canary Islands
  - H. Dr. José Molina Orrosos, Lanzarote, Canary Islands
  - H. Candelaria, Santa Cruz de Tenerife, Canary Islands
  - H. Dr. Negrín, Santa Cruz de Tenerife, Canary Islands
  - H. Universitario de Tenerife, Santa Cruz de Tenerife, Canary Islands
  - H. de Valdecilla, Santander, Cantabria
  - H. de León, León, Castille and León
  - H. Comarcal el Bierzo, Ponferrada, Castille and León
  - H. Clínico de Salamanca, Salamanca, Castille and León
  - H. Clinico de Valladolid, Valladolid, Castille and León
  - H. Río Ortega, Valladolid, Castille and León
  - H. de Albacete, Albacete, Castille-La Mancha
  - H. Ciudad Real, Ciudad Real, Castille-La Mancha
  - H. de Cuenca, Cuenca, Castille-La Mancha
  - H. de Manzanares, Manzanares, Castille-La Mancha
  - H. Alcázar, Toledo, Castille-La Mancha
  - H. Vírgen de la Salud, Toledo, Castille-La Mancha
  - H, de Tomelloso, Tomelloso, Castille-La Mancha
  - H. de Valdepeñas, Valdepeñas, Castille-La Mancha
  - H. Germans Trias Pujol, Badalona, Catalonia
  - H. Clínic, Barcelona, Catalonia
  - H. Sant Boi, Barcelona, Catalonia
  - H. Sant Pau, Barcelona, Catalonia
  - Hospital de Bellvitge, Barcelona, Catalonia
  - Xarxa Sanitaria i Social de Santa Tecla (Tarragona), El Vendrell, Catalonia
  - H. de Figueres, Figueres, Catalonia
  - H. Josep Trueta, Girona, Catalonia
  - H. Santa Caterina, Girona, Catalonia
  - H. General de Igualada, Igualada, Catalonia
  - H. Sant Joan de Déu de Manresa, Manresa, Catalonia
  - H. Sant Joan de Déu de Martorell, Martorell, Catalonia
  - H. Sant Joan de Reus, Reus, Catalonia
  - H. Parc Taulí de Sabadell, Sabadell, Catalonia
  - H. Esperit Sant, Santa Coloma de Gramanet, Catalonia
  - H. Joan XXIII, Tarragona, Catalonia
  - H. Verge de la Cinta de Tortosa, Tortosa, Catalonia
  - H. General de Vic, Vic, Catalonia
  - H. de Viladecans, Viladecans, Catalonia
  - H. Infanta Cristina, Badajoz, Extremadura
  - H. San Pedro Alcántara, Cáceres, Extremadura
  - H. de Coria/Plasencia, Coria, Extremadura
  - H. de Mérida, Mérida, Extremadura
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - H. Arquitecto Marcide, Ferrol, Galicia
  - Complexo Hospitalario Ourense, Ourense, Galicia
  - Complexo Hospitalario Pontevedra, Pontevedra, Galicia
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, Galicia
  - Complejo hospitalario Vigo, Vigo, Galicia
  - H. Meixoeiro, Vigo, Galicia
  - H. Xeral Cíes, Vigo, Galicia
  - POVISA, Vigo, Galicia
  - H. Puerta del Hierro, Madrid, Madrid
  - H. Santa Mª del Rosell, Cartagena, Murcia
  - H. de Arritxaca, El Palmar, Murcia
  - H. de Lorca, Lorca, Murcia
  - H. General de Múrcia, Murcia, Murcia
  - H. Morales Messeguer, Murcia, Murcia
  - H. de Navarra, Pamplona, Navarre
  - H. Central de Astúrias, Oviedo, Principality of Asturias
  - H. Vírgen del Rocío, Seville, Sevilla